CLINICAL TRIAL: NCT02891915
Title: A Phase IV Double-Blind, Placebo-Controlled, Randomized Trial to Evaluate Short Course vs.Standard Course Outpatient Therapy of Community Acquired Pneumonia in Children (SCOUT-CAP)
Brief Title: Trial to Evaluate Beta-Lactam Antimicrobial Therapy of Community Acquired Pneumonia in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-0079; HHSN272201300023I
Record Dates: First submitted 2016-09-01; First posted 2016-09-08 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2017-04-05

CONDITIONS: Pneumonia
Keywords: Antimicrobial; Beta-Lactam; Pneumonia; Short Course; Standard Course; Therapy
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin; Amoxicillin-Potassium Clavulanate Combination; Cefdinir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short (Active Comparator): 200 subjects will receive a short course of the initially prescribed antibiotic for 5 days plus 5 days of matching placebo
  Interventions: Drug: Amoxicillin; Drug: Amoxicillin-clavulanate; Drug: Cefdinir; Other: Placebo
- Standard (Active Comparator): 200 subjects will receive a standard course of the initially prescribed antibiotic( Amoxicillin, Amoxicillin-Clavulanate, Cefdinir) for 10 days
  Interventions: Drug: Amoxicillin; Drug: Amoxicillin-clavulanate; Drug: Cefdinir

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin is an aminopenicillin antibiotic
Drug: Amoxicillin-clavulanate — A fixed-ratio combination of amoxicillin trihydrate, an aminopenicillin, and potassium clavulanate, a beta-lactamase inhibitor, used to treat a broad-spectrum of bacterial infections, especially resistant strains.
Drug: Cefdinir — Cefdinir is a cephalosporin antibiotic used to treat bacterial infections in many different parts of the body.
Other: Placebo — Placebo
  Arms: Short

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, superiority clinical trial will test the effectiveness of short (5-day) vs.standard (10-day) course therapy in children who are diagnosed with CAP and initially treated in outpatient clinics, urgent care facilities, and emergency departments. Primary objective is to compare the composite overall outcome (Desirability of Outcome Ranking, DOOR) among children 6-71 months of age with CAP assigned to a strategy of short course (5 days) vs standard course (10 days) outpatient beta-lactam therapy at Outcome Assessment Visit #1 (Study Day 8 +/- 2 days)

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, superiority clinical trial evaluating short course (5 day) vs. standard course (10 day) of oral beta-lactam antibiotic therapy (amoxicillin, amoxicillin-clavulanate, cefdinir) for treatment of CAP in children 6-71 months of age who have clinically improved prior to enrollment. The study will randomize approximately 400 enrolled subjects to one of the two study arms (approximately 200 children in each arm) in order to reach 360 subjects completing Outcome Assessment Visit 1. Subjects will be randomized (1:1) to receive either a standard course of the initially prescribed antibiotic (10 days) or a short course of the initially prescribed antibiotic (5 days) plus 5 days of matching placebo. The study will recruit potential subjects from children who are diagnosed with CAP and who are initiated on oral beta-lactam therapy by healthcare providers in EDs, outpatient clinics, and urgent care centers at the study sites. Day -5 is defined as the date on which oral beta-lactam therapy is initiated for a diagnosis of CAP. Potential subjects will be identified at any time following clinical diagnosis of pneumonia. These subjects will be assessed for eligibility and enrolled on Day -3 to -1 of their initially prescribed oral beta-lactam therapy. Subjects may also be enrolled on Day 1 (the first day of receipt of study agent) provided they have not yet received any doses of the healthcare provider-prescribed antibiotic therapy for that day. The Primary objective is to compare the composite overall outcome (Desirability of Outcome Ranking, DOOR) among children 6-71 months of age with CAP assigned to a strategy of short course (5 days) vs standard course (10 days) outpatient beta-lactam therapy at Outcome Assessment Visit #1 (Study Day 8 +/- 2 days). The Secondary objectives are: 1) To compare the composite overall outcome (DOOR) among children 6-71 months of age with CAP assigned to a strategy of short course (5 days) vs standard course (10 days) outpatient beta-lactam therapy at Outcome Assessment Visit #2 (Study Day 22 +/- 3 days); 2) To compare the resolution of symptoms (a component of DOOR) among children 6-71 months of age with CAP assigned to a strategy of short course (5 days) vs standard course (10 days) outpatient beta-lactam therapy at Outcome Assessment Visits #1 and #2; 3) To compare the clinical response (a component of DOOR) among children 6-71 months of age with CAP assigned to a strategy of short course (5 days) vs standard course (10 days) outpatient beta-lactam therapy at Outcome Assessment Visits #1 and #2; 4) To compare solicited events (a component of DOOR) among children 6-71 months of age with CAP assigned to a strategy of short course (5 days) vs standard course (10 days) outpatient beta-lactam therapy at Outcome Assessment Visits #1 and #2; 5) To compare medically attended visits to Emergency Departments (ED) or outpatient clinics, hospitalizations, surgical procedures, and receipt of non-study systemic antibiotics (components of the clinical response) among children 6-71 months of age with CAP assigned to a strategy of short course (5 days) vs standard course (10 days) outpatient beta-lactam therapy at Outcome Assessment Visits #1 and #2

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 - 71 months
2. Provider diagnosis of CAP and prescription of antibiotic therapy with amoxicillin, amoxicillin-clavulanate, or cefdinir

   - amoxicillin or amoxicillin-clavulanate prescribed at a amoxicillin dose of 60 mg/kg/day

   -- cefdinir prescribed at a minimum dose of 10 mg/kg/day
3. Parental report of clinical improvement

   - based on lack of either subjective or known fever temperature >/= 38.3°C in the preceding 24 hours; current respiratory rate no greater than 50 breaths/minute (<2 years of age) or breaths/minute (= / > 2 years of age); and current grade of cough < 3
4. Ability of a parent or guardian to understand and comply with the study procedures and be available for all study visits
5. Signed written informed consent by a parent or guardian

Exclusion Criteria:

1. Treatment with any systemic antibiotic therapy within 7 days before the diagnosis of CAP 2. Initial therapy for CAP with combination antibiotic therapy

* amoxicillin, amoxicillin/clavulanate or cefdinir plus one or more additional oral, intravenous, or intramuscular antibiotics 3. History of anaphylaxis or severe drug allergy to amoxicillin, if prescribed amoxicillin or amoxicillin/clavulanic acid; or oral cephalosporin antibiotics (except cefaclor), if prescribed cefdinir 4. Presence of concomitant bacterial infection that requires > 5 days of antibiotic therapy 5. Radiographic findings (where applicable) of complicated pneumonia at presentation or any subsequent chest radiograph up to the time of enrollment
* clinically significant pleural effusion, lung abscess, or pneumatocele 6. Hospitalization for pneumonia during Day -5 to -1 of antibiotic therapy for CAP
* subjects who require serial clinical assessments, but are discharged within 24 hours will not be considered hospitalized and will not satisfy this exclusion criterion 7. Pneumonia due to S. aureus or group A streptococcus documented by positive blood culture or PCR, at the time of enrollment 8. History of pneumonia within the previous 6 months 9. History of persistent asthma within the previous 6 months or current acute asthma exacerbation
* persistent asthma is defined as receiving daily asthma maintenance therapy such as inhaled corticosteroids, cromolyn, theophylline, or leukotriene receptor antagonists

  -- acute asthma exacerbation is defined as receiving concomitant bronchodilator therapy and systemic corticosteroids 10. Provider-diagnosis of aspiration pneumonia, bronchiolitis, or bronchitis 11. Surgery or other invasive procedures of the upper or lower airway (e.g., bronchoscopy, laryngoscopy) with general anesthesia or hospitalization </=7 days before diagnosis of CAP 12. History of an underlying chronic medical condition
* including chronic heart disease, chronic lung disease (except asthma), congenital anomalies of the airways or lung, cystic fibrosis, chronic renal disease including nephrotic syndrome, protein-losing enteropathy of any cause, severe malnutrition, neurocognitive disorders, metabolic disorders (including phenylketonuria), or genetic disorders (note: genetic syndromes such as Down syndrome and Edwards Syndrome are excluded; however, children with genetic disorders (e.g., hemophilia) but who do not have a genetic syndrome may not satisfy this particular exclusion criterion; it is important that children with such genetic disorders do not have symptoms and/or comorbidities that would pose additional risk to them nor jeopardize the adequacy of study assessments.) 13. History of a condition that compromises the immune system
* HIV infection, primary immunodeficiency, anatomic or functional asplenia; receipt of a hematopoietic stem cell or solid organ transplant at any time; receipt of immunosuppressive therapy including chemotherapeutic agents, biologic agents, antimetabolites or radiation therapy during the past 12 months; or daily use of systemic corticosteroids for more than 7 consecutive days during the past 14 days 14. Any other condition that in the judgment of the investigator precludes participation because it could affect the safety of the subject 15. Current enrollment in another clinical trial of an investigational agent 16. Previous enrollment in this trial

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 385 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Alabama - Children's of Alabama - Infectious Diseases/Virology, Birmingham, Alabama
  - Arkansas Children's Hospital - Infectious Diseases, Little Rock, Arkansas
  - University of Louisville School of Medicine - Norton Children's Hospital - Infectious Diseases, Louisville, Kentucky
  - Washington University School of Medicine in St. Louis - Infectious Diseases, St Louis, Missouri
  - Duke Human Vaccine Institute - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Children's Hospital of Philadelphia - The Center for Pediatric Clinical Effectiveness, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC - General Academic Pediatric, Pittsburgh, Pennsylvania
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee

REFERENCES:
- [Derived] Pettigrew MM, Kwon J, Gent JF, Kong Y, Wade M, Williams DJ, Creech CB, Evans S, Pan Q, Walter EB, Martin JM, Gerber JS, Newland JG, Hofto ME, Staat MA, Fowler VG, Chambers HF, Huskins WC; Antibacterial Resistance Leadership Group. Comparison of the Respiratory Resistomes and Microbiota in Children Receiving Short versus Standard Course Treatment for Community-Acquired Pneumonia. mBio. 2022 Apr 26;13(2):e0019522. doi: 10.1128/mbio.00195-22. Epub 2022 Mar 24. PMID 35323040
- [Derived] Williams DJ, Creech CB, Walter EB, Martin JM, Gerber JS, Newland JG, Howard L, Hofto ME, Staat MA, Oler RE, Tuyishimire B, Conrad TM, Lee MS, Ghazaryan V, Pettigrew MM, Fowler VG Jr, Chambers HF, Zaoutis TE, Evans S, Huskins WC; The DMID 14-0079 Study Team. Short- vs Standard-Course Outpatient Antibiotic Therapy for Community-Acquired Pneumonia in Children: The SCOUT-CAP Randomized Clinical Trial. JAMA Pediatr. 2022 Mar 1;176(3):253-261. doi: 10.1001/jamapediatrics.2021.5547. PMID 35040920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children, males and females, aged 6-71 months who are diagnosed with Community Acquired Pneumonia (CAP) and initially treated in outpatient clinics, urgent care facilities, and emergency departments were enrolled. Participants were enrolled between 02DEC2016 and 22NOV2019.
Groups:
- Short Course: Participants will receive a short course of the initially prescribed antibiotic for 5 days plus 5 days of matching placebo
  Amoxicillin: Amoxicillin is an aminopenicillin antibiotic
  Amoxicillin-clavulanate: A fixed-ratio combination of amoxicillin trihydrate, an aminopenicillin, and potassium clavulanate, a beta-lactamase inhibitor, used to treat a broad-spectrum of bacterial infections, especially resistant strains.
  Cefdinir: Cefdinir is a cephalosporin antibiotic used to treat bacterial infections in many different parts of the body.
  Placebo: Placebo
- Standard Course: Participants will receive a standard course of the initially prescribed antibiotic (Amoxicillin, Amoxicillin-Clavulanate, Cefdinir) for 10 days
  Amoxicillin: Amoxicillin is an aminopenicillin antibiotic
  Amoxicillin-clavulanate: A fixed-ratio combination of amoxicillin trihydrate, an aminopenicillin, and potassium clavulanate, a beta-lactamase inhibitor, used to treat a broad-spectrum of bacterial infections, especially resistant strains.
  Cefdinir: Cefdinir is a cephalosporin antibiotic used to treat bacterial infections in many different parts of the body.
Period: Overall Study
Arm/Group | Short Course | Standard Course
Started | 192 | 193
Completed | 179 | 181
Not Completed | 13 | 12
Not completed — Enrolled but Treatment Not Administered | 6 | 4
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Became Ineligible After Enrollment | 2 | 1
Not completed — Lost to Follow-up | 1 | 4
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Course: Participants will receive a standard course of the initially prescribed antibiotic( Amoxicillin, Amoxicillin-Clavulanate, Cefdinir) for 10 days
  Amoxicillin: Amoxicillin is an aminopenicillin antibiotic
  Amoxicillin-clavulanate: A fixed-ratio combination of amoxicillin trihydrate, an aminopenicillin, and potassium clavulanate, a beta-lactamase inhibitor, used to treat a broad-spectrum of bacterial infections, especially resistant strains.
  Cefdinir: Cefdinir is a cephalosporin antibiotic used to treat bacterial infections in many different parts of the body.
- Total: Total of all reporting groups
Arm/Group | Short Course | Standard Course | Total
Number analyzed (Participants) | 192 | 193 | 385
Age, Continuous [Mean (Standard Deviation); unit: months] | 34.6 (16.6) | 36.8 (17.8) | 35.7 (17.2)
Age, Customized [Count of Participants; unit: Participants]
  < 24 Months | 55 | 56 | 111
  24-71 Months | 137 | 137 | 274
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 93 | 190
  Male | 95 | 100 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 18 | 33
  Not Hispanic or Latino | 176 | 173 | 349
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 48 | 51 | 99
  White | 121 | 118 | 239
  More than one race | 15 | 17 | 32
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 192 | 193 | 385
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Arkansas Children's Hospital | 8 | 5 | 13
  United States: Children's Hospital of Philadelphia | 59 | 63 | 122
  United States: Children's Hospital of Pittsburgh | 67 | 62 | 129
  United States: Cincinnati Children's Hospital | 2 | 2 | 4
  United States: Duke University | 23 | 20 | 43
  United States: University of Alabama at Birmingham-Pediatrics | 1 | 6 | 7
  United States: Vanderbilt University Medical Center | 16 | 16 | 32
  United States: Washington University | 16 | 19 | 35
Initial Antibiotic [Count of Participants; unit: Participants]
  Amoxicillin | 176 | 174 | 350
  Amoxicillin Clavulanate | 10 | 10 | 20
  Cefdinir | 6 | 9 | 15
Initial Site of Treatment [Count of Participants; unit: Participants]
  ED | 41 | 40 | 81
  Out-Patient/Urgent Care | 151 | 153 | 304

OUTCOME MEASURES:

1. Primary Outcome: Desirability of Outcome Ranking (DOOR)
Description: DOOR is a composite endpoint created using clinical outcomes from the first 5 days and at Outcome Assessment Visit #1 (OAV #1). It is based on adequate clinical response at OAV #1, solicited symptoms from first 5 days and number of days of antibiotics use for worsening pneumonia from the first 5 days of the study.
Time Frame: Outcome Assessment Visit 1 (Study Day 8 +/- 2 days)
Population: Intent to Treat (ITT) Population: All randomized subjects that were still eligible on Day 1 of the study. Analysis of DOOR will use all subjects in the ITT population. Subjects with missing values of DOOR will have their values imputed. However, summaries of observed ordinal clinical response values presented below are based on complete data without imputation.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 170 | 174
Participants
  Adequate clinical response with resolution of symptoms and no adverse events | 97 | 107
  Adequate clinical response with resolution of symptoms and with mild adverse events | 47 | 42
  Adequate clinical response with resolution of symptoms and with moderate adverse events | 14 | 10
  Adequate clinical response with resolution of symptoms and with severe adverse events | 0 | 2
  Adequate clinical response with persistent symptoms of fever, tachypnea, or cough | 10 | 12
  Lack of adequate clinical response with ED/clinic visit but no hospitalization | 2 | 1
  Lack of adequate clinical response with hospitalization | 0 | 0
  Death from any cause | 0 | 0
Statistical Analysis 1: Comparison: Short Course vs Standard Course; Null: the sum of the probability that a subject assigned to the 5-day arm will have a higher DOOR (higher DOOR is a lower value and is superior) than if assigned to the 10-day arm plus one-half the probability of equal DOORs is 50% (i.e., no difference in DOOR); Test type: Superiority — DOOR is a composite endpoint created using clinical outcomes from the first 5 days and at Outcome Assessment Visit #1 (OAV #1). It is based on adequate clinical response at OAV #1, solicited symptoms from first 5 days and number of days of antibiotics use for worsening pneumonia from the first 5 days of the study; p < 0.001, Wilcoxon (Mann-Whitney) — Missing DOOR values at OAV #1 were first imputed using linear regression using baseline covariates and available DOOR components as covariates; The Mann-Whitney test was run on the multiple imputed datasets to generate estimates of DOOR probability and p-value; Pr (Higher DOOR in Short-Course) = 0.69, 95% CI 2-sided [0.63 to 0.75]

2. Secondary Outcome: Desirability of Outcome Ranking (DOOR)
Description: DOOR is a composite endpoint created using clinical outcomes from the first 18 days and at Outcome Assessment Visit #2 (OAV #2). It is based on adequate clinical response at OAV #2, solicited symptoms from first 18 days and number of days of antibiotics use for worsening pneumonia from the first 18 days of the study.
Time Frame: Outcome Assessment Visit 2 (Study Day 22 +/- 3 days)
Population: ITT Population: All randomized subjects that were still eligible on Day 1 of the study. Analysis of DOOR will use all subjects in the ITT population. Subjects with missing values of DOOR will have their values imputed. However, summaries of observed ordinal clinical response values presented below are based on complete data without imputation.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 163 | 167
Participants
  Adequate clinical response with resolution of symptoms and no solicited events | 73 | 81
  Adequate clinical response with resolution of symptoms and with mild solicited events | 53 | 51
  Adequate clinical response with resolution of symptoms and with moderate solicited events | 25 | 20
  Adequate clinical response with resolution of symptoms and with severe solicited events | 3 | 4
  Adequate clinical response with persistent symptoms of fever, tachypnea, or cough | 7 | 8
  Lack of adequate clinical response with ED/clinic visit but no hospitalization | 2 | 3
  Lack of adequate clinical response with hospitalization | 0 | 0
  Death from any cause | 0 | 0
Statistical Analysis 1: Comparison: Short Course vs Standard Course; Null: the sum of the probability that a subject assigned to the 5-day arm will have a higher DOOR (higher DOOR is a lower numerical value and is superior) than if assigned to the 10-day arm plus one-half the probability of equal DOORs is 50% (i.e., no difference in DOOR); Test type: Superiority — Testing whether Short course is superior to Standard course based on DOOR at OAV #2; p < 0.001, Wilcoxon (Mann-Whitney) — Missing DOOR values at OAV #2 were first imputed using linear regression using baseline covariates and available DOOR components as covariates; The Mann-Whitney test was run on the multiple imputed datasets to generate estimates of DOOR probability and p-value; Pr (Higher DOOR in Short-Course) = 0.63, 95% CI 2-sided [0.57 to 0.69]

3. Secondary Outcome: Resolution of Symptoms (a Component of DOOR)
Description: This table provides number and percentage of subjects who experienced lack of resolution of symptoms by their OAV #1.
Time Frame: Outcome Assessment Visit 1 (Study Day 8 +/- 2 days)
Population: Complete Case at OAV #1. This population is made of subjects who were treated with at least one dose of study product, did not terminate early from the study before OAV #1, and completed OAV #1 with non-missing data for all DOOR components at OAV #1.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 170 | 174
Participants
  Lack of Resolution of Symptoms | 12 | 13
  Fever | 2 | 1
  Elevated respiratory rate | 2 | 7
  Cough | 7 | 4

4. Secondary Outcome: Resolution of Symptoms (a Component of DOOR)
Description: This table provides number and percentage of subjects who experienced lack of resolution of symptoms by their OAV #2.
Time Frame: Outcome Assessment Visit 2 (Study Day 22 +/- 3 days)
Population: Complete Case at OAV #2. This population is made of subjects who were treated with at least one dose of study product, did not terminate early from the study before OAV #2, and completed OAV #2 with non-missing data for all DOOR components at OAV #2.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 163 | 167
Participants
  Lack of Resolution of Symptoms | 9 | 11
  Fever | 0 | 3
  Elevated respiratory rate | 2 | 1
  Cough | 6 | 5

5. Secondary Outcome: Adequate Clinical Response Rates (a Component of DOOR)
Description: Lack of adequate clinical response at OAV #1 is defined as the presence of a medically attended visit to an Emergency Department (ED) or outpatient clinic or hospitalization or receipt of non-study antibiotics or surgical procedures for persistent or worsening pneumonia from Day 1 to Day 5.
Time Frame: Outcome Assessment Visit 1 (Study Day 8 +/- 2 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 170 | 174
Participants
  Lack of Adequate Clinical Response | 2 | 1
  ED or Clinic Visit | 2 | 1
  Receipt of Non-Study Antibiotic | 2 | 1
  Hospitalization | 0 | 0
  Surgical Procedure | 0 | 0

6. Secondary Outcome: Adequate Clinical Response Rates (a Component of DOOR)
Description: Lack of adequate clinical response at OAV #2 is defined as the presence of a medically attended visit to an ED or outpatient clinic or hospitalization or receipt of non-study antibiotics or surgical procedures for persistent or worsening pneumonia from Day 1 to Day 18.
Time Frame: Outcome Assessment Visit 2 (Study Day 22 +/- 3 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 163 | 167
Participants
  Lack of Adequate Clinical Response | 2 | 3
  ED or Clinic Visit | 4 | 2
  Receipt of Non-Study Antibiotic | 2 | 3
  Hospitalization | 0 | 0
  Surgical Procedure | 0 | 0

7. Secondary Outcome: Number of Participants Reporting Solicited Symptoms
Description: This table summarizes the number and percentage of subjects experiencing any solicited events of mild, moderate or severe severity from Day 1 to Day 5
Time Frame: Outcome Assessment Visit 1 (Study Day 8 +/- 2 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 170 | 174
Participants
  Any Event | 74 | 68
  Irritability | 52 | 43
  Vomiting | 11 | 11
  Diarrhea | 23 | 21
  Allergic Reaction | 15 | 15
  Stomatitis | 1 | 3
  Candidiasis | 4 | 4

8. Secondary Outcome: Number of Participants Reporting Solicited Symptoms
Description: This table summarizes the number and percentage of subjects experiencing any solicited events of mild, moderate or severe severity from Day 1 to Day 18
Time Frame: Outcome Assessment Visit 2 (Study Day 22 +/- 3 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 163 | 167
Participants
  Any Event | 91 | 89
  Irritability | 67 | 60
  Vomiting | 19 | 24
  Diarrhea | 33 | 30
  Allergic Reaction | 22 | 21
  Stomatitis | 1 | 6
  Candidiasis | 7 | 7

9. Secondary Outcome: Number of Participants Receiving Non-study Systemic Antibiotics for Persistent or Worsening Pneumonia During Medically Attended Visits
Description: This table provides number and percentage of subjects who received non-study antibiotics for any use from Day 1 to Day 5
Time Frame: Outcome Assessment Visit 1 (Study Day 8 +/- 2 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 170 | 174
Participants
  ED or Clinic Visit | 2 | 1
  Receipt of Non-Study Antibiotic | 2 | 1

10. Secondary Outcome: Number of Participants Receiving Non-study Systemic Antibiotics for Persistent or Worsening Pneumonia During Medically Attended Visits
Description: This table provides number and percentage of subjects who received non-study antibiotics for any use from Day 1 to Day 18
Time Frame: Outcome Assessment Visit 2 (Study Day 22 +/- 3 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 163 | 167
Participants
  ED or Clinic Visit | 4 | 2
  Receipt of Non-Study Antibiotic | 2 | 3

11. Secondary Outcome: Number of Participants Receiving Non-study Systemic Antibiotics for All Causes During Medically Attended Visits
Description: This table provides number and percentage of subjects who received non-study antibiotics for any reason from Day 1 to Day 5
Time Frame: Outcome Assessment Visit 1 (Study Day 8 +/- 2 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 170 | 174
Participants
  ED or Clinic Visit | 8 | 7
  Receipt of Non-Study Antibiotic | 7 | 2

12. Secondary Outcome: Number of Participants Receiving Non-study Systemic Antibiotics for All Causes During Medically Attended Visits
Description: This table provides number and percentage of subjects who received non-study antibiotics for any reason from Day 1 to Day 18
Time Frame: Outcome Assessment Visit 2 (Study Day 22 +/- 3 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Standard Course
Number analyzed (Participants) | 163 | 167
Participants
  ED or Clinic Visit | 29 | 32
  Receipt of Non-Study Antibiotic | 18 | 11

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred from Receipt of Study Agent (Day 1) through the final Outcome Assessment Visit (Day 22 +/- 3 days) were reported.
Description: Solicited AEs for both the Short and Standard course were assessed using MedDRA 22.0.
Arm/Group | Short Course | Standard Course
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/193
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/193
Other Adverse Events (participants affected / at risk) | 98/192 | 98/193
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Course (N=192) | Standard Course (N=193)
Irritability (General disorders) | 73 (370) | 65 (313)
Vomiting (Gastrointestinal disorders) | 23 (41) | 28 (62)
Diarrhea (Gastrointestinal disorders) | 37 (124) | 34 (125)
Allergic Reaction (Immune system disorders) | 22 (98) | 23 (156)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT02891915/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT02891915/SAP_001.pdf